CLINICAL TRIAL: NCT07390292
Title: The Effect of Cognitive Functions on Functional Capacity, Balance, Fear of Falling and Quality of Life in Patients With Type 2 Diabetes
Brief Title: Assessment of Cognitive Function and Functional Performance in Patients With Type 2 Diabetes
Status: Not yet recruiting | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025/251
Record Dates: First submitted 2026-01-05; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes Mellitus; Cognitive Function; Balance; Functional Capacity
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Type 2 Diabetes Mellitus Group
  Interventions: Other: No intervention (observational study)
- Healthy Control Group
  Interventions: Other: No intervention (observational study)

INTERVENTIONS:
Other: No intervention (observational study) — This is an observational study. No treatment was applied to the individuals. The study will evaluate the individuals' cognitive functions and functional capacities, balance, fear of falling, and quality of life.

SUMMARY:
Diabetes is a chronic metabolic disease that is becoming a growing public health problem worldwide, affecting people's lives in many ways. It is characterized by impaired carbohydrate, lipid, and protein metabolism associated with insufficient insulin secretion and/or reduced sensitivity to the metabolic effects of insulin.Along with diabetes, many complications may develop in affected individuals. Cognitive impairments are now also considered an important and common complication of diabetes.The aim of this study is to investigate the effects of cognitive function levels on functional capacity, balance, fear of falling, and quality of life in individuals with type 2 diabetes.In this context, participants' cognitive function levels will be assessed using the Mini-Mental State Examination and the Stroop Test. Functional capacity will be evaluated using the 6-Minute Walk Test. Balance performance will be assessed using the Biodex Balance System and the Four Square Step Test. Lower extremity muscle strength will be measured using a digital hand-held dynamometer and the 30-Second Sit-to-Stand Test. Fear of falling will be evaluated using the Falls Efficacy Scale-International (FES-I), the Functional Reach Test, and the Timed Up and Go (TUG) Test. Participants' quality of life will be assessed using the WHOQOL-BREF quality of life questionnaire.

DETAILED DESCRIPTION:
The study will include 40 volunteer patients diagnosed with Type 2 Diabetes Mellitus and a control group consisting of 40 healthy individuals without any chronic disease, matched in terms of age and sex. The research will be conducted at the Cardiac and Pulmonary Physiotherapy and Physiotherapy and Rehabilitation Education and Research Laboratory of Bezmialem Vakıf University Eyüp Campus. This study is designed as a cross-sectional study based on the objective evaluation of the current condition without any intervention or treatment.

Written informed consent will be obtained from all participants prior to participation. Subsequently, the demographic and clinical data of the participants will be recorded. Cognitive functions will be assessed using the Mini-Mental State Examination (MMSE) and the Stroop Test. Body composition will be measured using the digital and portable Omron BF511 Body Composition Monitor. Lower extremity muscle strength will be evaluated using an electronic hand-held dynamometer, and in addition, the 30-Second Sit-to-Stand Test will be performed.

Balance performance will be assessed using the Biodex Balance System; within this system, the Postural Stability Test, Limits of Stability Test, and Sensory Organization Test will be performed. In addition, the Four Square Step Test will also be conducted as a measure to support the assessment of dynamic balance.

Fear of falling will be assessed using the Falls Efficacy Scale-International (FES-I), the Functional Reach Test, and the Timed Up and Go (TUG) Test. Participants' quality of life levels will be determined using the WHOQOL-BREF Quality of Life Questionnaire. All obtained results will be compared between individuals with type 2 diabetes and the healthy control group; the relationships between cognitive function levels and functional capacity, balance, fear of falling, and quality of life will be examined using statistical analyses.

The implementation of all assessments takes approximately 40-45 minutes for each participant.

Statistical analysis of the data will be performed using SPSS v.20 software, and a significance level of p<0.05 will be accepted.

ELIGIBILITY:
Inclusion Criteria:

* Being between 40 and 65 years of age
* Having an HbA1c level between 6.5 and 11
* Having been diagnosed with diabetes for at least 1 year
* Scoring 24 or higher on the Mini-Mental State Examination
* Being able to walk independently without assistance
* Having provided voluntary participation and signed written informed consent

Exclusion Criteria:

* Having a diagnosis of any neurological or psychiatric disorder (e.g., hemiplegia, Alzheimer's disease, Parkinson's disease)
* Having uncontrolled hypertension and/or uncontrolled cardiac arrhythmia
* Having vertigo or other vestibular system disorders
* Having major musculoskeletal disorders
* Having undergone percutaneous transluminal coronary angioplasty or having a cardiac pacemaker
* Being pregnant
* Being unable to read or write in Turkish

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be conducted at Bezmialem Vakif University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, including the Pulmonary Physiotherapy and Rehabilitation Education and Research Laboratory and the Cardiac Physiotherapy and Rehabilitation Education and Research Laboratory, using face-to-face interview methods with the participants.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Postural Stability | Single assessment at baseline
  Postural stability will be assessed using the Biodex Balance System®. This assessment is performed to evaluate the individual's ability to maintain the center of body mass.
  Deviations from the center of balance will be recorded during the test. Higher stability index scores indicate greater deviation from the center of balance and poorer postural stability.
Limits of Stability | Single assessment at baseline
  This assessment will be conducted using the Biodex Balance System®. The test will be performed on a static platform. The purpose of the test is to evaluate the individual's ability to shift and control the center of body mass within the base of support.
  Directional control (overall, forward, backward, left, right, forward/left, forward/right, backward/left, backward/right) will be assessed and expressed as a percentage (%).
  Higher scores are associated with better postural control.
Sensory Integration of Balance | Single assessment at baseline
  This assessment will be conducted using the Biodex Balance System®. The purpose of the test is to evaluate how different sensory inputs contribute to the maintenance of balance and how well balance can be preserved when one or more of these sensory inputs are removed.
  The test will be performed under the following conditions: eyes open and eyes closed on a firm surface, and eyes open and eyes closed on a foam surface.
  A sway index will be calculated for each condition.

SECONDARY OUTCOMES:
Stroop Test | Single assessment at baseline
  The Stroop Test is used to assess cognitive function, including processing speed, selective attention, cognitive flexibility, and the ability to inhibit automatic responses.The test consists of three parts, in which participants are required to perform color-word tasks. The completion time of the test will be recorded in seconds.
Mini-Mental State Examination (MMSE) | Single assessment at baseline
  The Mini-Mental State Examination (MMSE) will be used to assess general cognitive function. The test evaluates the domains of orientation, attention, memory, calculation, and language. The total score ranges from 0 to 30, with higher scores indicating better cognitive performance.
Four Square Step Test | Single assessment at baseline
  It is used to assess dynamic balance during obstacle negotiation. The patient is instructed to step over four canes placed on the floor in a cross configuration, following a specified sequence.
  The completion time of the test is recorded in seconds.
Assessment of Functional Capacity | Single assessment at baseline
  Functional capacity will be assessed using the 6-minute walk test. This test involves participants walking along a 30-meter corridor at their own pace for six minutes, with the distance recorded in meters. At the end of six minutes, the participant is informed that the test is complete and the test is terminated. The expected average walking distance for healthy individuals ranges from 400 to 700 meters.
30 Second Sit to Stand Test | Single assessment at baseline
  Lower extremity muscle strength will be assessed using the 30-second chair stand test.
  During the test, participants will be instructed to stand up from a chair for 30 seconds with their arms crossed over their chest and their feet flat on the floor.
  The number of completed stands will be recorded to evaluate functional lower extremity muscle strength.
Quadriceps Femoris Muscle Strength | Single assessment at baseline
  Quadriceps femoris muscle strength will be assessed using an electronic hand-held dynamometer.Participants will be instructed to sit with the knee in full extension, while the physiotherapist applies maximal resistance at the ankle to evaluate the isometric strength of the quadriceps femoris muscle.The muscle strength value will be recorded in kilograms (kg).
Falls Efficacy Scale-International (FES-I) | Single assessment at baseline
  To assess fear of falling, fear of falling will be assessed using the Falls Efficacy Scale-International (FES-I).The scale consists of 16 items that assess individuals' levels of concern related to falling during daily activities.Each item is scored from 1 (not at all concerned) to 4 (very concerned).
  The total score will be recorded.
Functional Reach Test | Single assessment at baseline
  The Functional Reach Test is performed to assess fall risk. During the test, participants are instructed to stand, raise the arm to approximately 90 degrees, and reach forward as far as possible without stepping or losing balance.The distance between the starting position of the hand and the furthest point reached is recorded in centimeters (cm).Values of 15 cm or less indicate an increased risk of falling.
Timed Up and Go (TUG) Test | Single assessment at baseline
  The Timed Up and Go (TUG) Test is performed to assess fall risk. The test requires a chair and a stopwatch. A 3-meter distance is marked in front of the chair, and participants are instructed to stand up from the chair on the command "go," walk this distance at a normal pace, and sit down again.
  The completion time of the test is recorded in seconds. Longer completion times are associated with an increased risk of falling.
Assessment of Quality of Life | Single assessment at baseline
  Quality of life will be assessed using the WHOQOL-BREF questionnaire. The WHOQOL-BREF consists of four domains: physical health (7 items), psychological well-being (6 items), social relationships (3 items), and environmental health (8 items). All items are rated on a 5-point Likert scale and scored from 1 to 5.
Body Mass İndex | Single assessment at baseline
  Body mass index will be taken into consideration during evaluation. Body height (m) will be measured using standardized procedures, and body weight (kg) will be measured using the Omron BF511 Body Composition Monitor. Body Mass Index (BMI) will be calculated by dividing body weight (kg) by the square of height in meters (kg/m²).
Body Fat Mass (kg) | Single assessment at baseline
  Body fat mass (kg) will be measured using the Omron BF511 Body Composition Monitor according to the standard protocol of the device.
Skeletal Muscle Mass (kg) | Single assessment at baseline
  Skeletal muscle mass (kg) will be measured using the Omron BF511 Body Composition Monitor according to the standard protocol of the device.
Resting Metabolic Rate | Single assessment at baseline
  Resting metabolic rate (kcal) will be assessed using the Omron BF511 Body Composition Monitor.
Visceral Fat Level | Single assessment at baseline
  Visceral fat level will be assessed using the Omron BF511 Body Composition Monitor according to the manufacturer's instructions.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)